CLINICAL TRIAL: NCT06961968
Title: A Multicenter, Double-Blind, Randomized Withdrawal Study in Patients With Schizophrenia Receiving Either Iloperidone Long-Acting Injection (LAI) or Placebo Injection
Brief Title: Randomized Withdrawal Study in Patients With Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VYV-683-3102
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic Agents; Iloperidone; Long-Acting Injection; Randomized Withdrawal
MeSH Terms: conditions — Schizophrenia | interventions — iloperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iloperidone (Experimental): During the 12-week stabilization phase, all patients will receive open-label iloperidone administered as oral tablets (weeks 1-6) and as long-acting intramuscular injections (weeks 7-12). Subsequently, patients will be randomized in a 1:1 ratio to one of two arms: iloperidone long-acting injection or matching placebo. Post-randomization this arm will receive double-blind study drug (iloperidone long-acting injection) as long-acting intramuscular injections for up to 52 weeks.
  Interventions: Drug: iloperidone
- placebo (Placebo Comparator): During the 12-week stabilization phase, all patients will receive open-label iloperidone administered as oral tablets (weeks 1-6) and as long-acting intramuscular injections (weeks 7-12). Subsequently, patients will be randomized in a 1:1 ratio to one of two arms: iloperidone long-acting injection or matching placebo. Post-randomization this arm will receive double-blind study drug (matching placebo) as long-acting intramuscular injections for up to 52 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: iloperidone — iloperidone LAI
  Arms: iloperidone
Drug: placebo — matching placebo
  Arms: placebo

SUMMARY:
The purpose of this research is to evaluate the efficacy of dosing iloperidone long-acting injection (LAI) compared to placebo in preventing the exacerbation of symptoms in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 to 65 years of age (inclusive)
* Diagnosed with schizophrenia per DSM-5 criteria
* In need of ongoing psychiatric treatment

Exclusion Criteria:

* DSM-5 diagnosis of a psychiatric disorder other than schizophrenia that was the primary focus of treatment within the previous six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Time to exacerbation of symptoms | Up to 52 weeks post-randomization
  As measured by the time to first exacerbation of psychiatric symptoms

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Vanda Investigational Site, Rogers, Arkansas
  - Vanda Investigational Site, Costa Mesa, California
  - Vanda Investigational Site, Lemon Grove, California
  - Vanda Investigational Site, Oceanside, California
  - Vanda Investigational Site, Pico Rivera, California
  - Vanda Investigational Site, San Diego, California
  - Vanda Investigational Site, Walnut Creek, California
  - Vanda Investigational Site, North Miami, Florida
  - Vanda Investigational Site, Atlanta, Georgia
  - Vanda Investigational Site, Peachtree Corners, Georgia
  - Vanda Investigational Site, Chicago, Illinois
  - Vanda Investigational Site, Flowood, Mississippi
  - Vanda Investigational Site, Saint Charles, Missouri
  - Vanda Investigational Site, St Louis, Missouri
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, Marlton, New Jersey
  - Vanda Investigational Site, Staten Island, New York
  - Vanda Investigational Site, Austin, Texas
  - Vanda Investigational Site, Houston, Texas
  - Vanda Investigational Site, Irving, Texas
  - Vanda Investigational Site, Richardson, Texas
  - Vanda Investigational Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No